CLINICAL TRIAL: NCT04250480
Title: Changes in Cognition During a 24-h Simulated Military Operation (SUSOP). Influence of β-alanine Supplementation and Markers of Classical Monocyte Recruitment
Brief Title: Changes in Cognition During a 24-h Simulated Military Operation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Collaborators: National Strength and Conditioning Association (Other)
Responsible Party: Principal Investigator, Adam Wells, Assistant Professor, University of Central Florida
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SBE-17-13223
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Cognitive Impairment
Keywords: beta-alanine; immune cells
MeSH Terms: conditions — Cognitive Dysfunction | interventions — beta-Alanine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta-alanine (Experimental): 4 g by mouth, 3 times per day with regular meals for 14 days.
  Interventions: Dietary Supplement: beta-alanine
- Placebo (Placebo Comparator): 4 g by mouth, 3 times per day with regular meals for 14 days.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: beta-alanine — beta-alanine tablet
  Arms: Beta-alanine
Dietary Supplement: placebo — rice powder tablet
  Arms: Placebo

SUMMARY:
Sustained military operations (SUSOPs) result in psychological stress and cognitive dysfunction, which may be related to the recruitment of classical monocytes into the brain.

Goals:

* To investigate the effect of sustained-release beta-alanine on changes in cognition and markers of immune cell recruitment during a 24-hour simulated military operation.
* To examine associations between changes cognition and changes in markers mediating immune cell recruitment.

DETAILED DESCRIPTION:
Sustained military operations (SUSOPs) expose soldiers to a multitude of stressors, including sustained physical activity, caloric deficit, and sleep deprivation. Several studies have shown that the combination of these factors result in psychological stress, which often leads to significant cognitive impairment.

Psychological stress has been shown to result in activation of neuroendocrine pathways that signal into the periphery and relay information from the brain to the immune system. This process is generally characterized by elevations of several key pro-inflammatory cytokines, chemokines, secondary messengers and reactive oxygen species. Notably, peripheral classical monocytes are reported to undergo recruitment to the brain during periods of psychological stress following priming by cytokines secreted from activated microglia.

Carnosine, an endogenous dipeptide consisting of beta-alanine and L-histidine, has been shown to inhibit the synthesis of inflammatory and oxidative mediators in microglia in vitro. Beta-alanine, which is the rate limiting amino acid in carnosine formation has been shown to increase carnosine concentrations in various regions of the brain in rodents which been associated with biochemical changes that resulted in favorable improvements in resilience to stress exposure. However, data on the effects of beta-alanine supplementation on cognition in humans is less clear. Further, the effect of beta-alanine supplementation on systemic and cellular mediators of monocyte recruitment has not been examined.

Goals:

* To investigate the effect of sustained-release beta-alanine on changes in psychological stress and cognition using Automated Neuropsychological Assessment Metric (ANAM) cognitive assessments during a 24-hour simulated military operation.
* To examine the effect of sustained-release beta-alanine on monocyte chemoattractant protein-1 (MCP-1), interleukin-8, Lymphocyte function-associated antigen-1 (CD11a), macrophage-1-antigen (CD11b) expression and C-C chemokine receptor 2 (CCR2) expression on neutrophils and classical monocytes during a 24-hour simulated military operation.
* To examine associations between MCP-1, interleukin-8, CD11a, CD11b, CCR2 and a composite measure of cognition derived from ANAM assessment scores during a 24-hour simulated military operation.

Method:

Double-blind placebo controlled trial compared the effect of supplementation with sustained release beta-alanine (12 grams per day) versus placebo (equivalent amount of rice powder) on cognition and monocyte responses during a 24-hour simulated military operation consisting of sleep-restriction, caloric restriction, and acute and sustained periods military specific physical activity.

Supplementation occurred over a period of 14 days prior to completion of the simulated military operation. ANAM tests were assessed and blood samples taken upon arrival to the lab for the 24 hour simulated operation (0 hours) and at 12, 18 and 24 hours during the SUSOP.

ELIGIBILITY:
Inclusion Criteria:

* Participants in this study will be males aged 18-35, preferably with military training or are current Reserve Officers' Training Corps cadets
* Free of any physical limitations (determined by medical and activity history questionnaire [MHQ] and the physical activity readiness questionnaire [PAR-Q+]).
* Participants will be required to be recreationally-active (defined according to American College of Sports Medicine standards of at least 150 minutes exercise per week).
* Participants must be willing abstain from dietary supplementation throughout the duration of the study.
* Participant understands the study procedures and signs forms providing informed consent to participate in the study.

Exclusion Criteria:

* Individual does not provide consent to participate in this study.
* Inability to perform physical exercise (determined by health and activity questionnaire [MHQ] and physical activity readiness questionnaire [PAR-Q+]). That is Answering "Yes" to any question on the PAR-Q+, or having a pre-existing condition such as musculoskeletal injury, back pain, chronic pain etc. that the investigative team perceives will prevent a participant from safely completing the protocol.
* Taking any other nutritional supplement or performance-enhancing drug (determined from health and activity questionnaire).
* Regularly taking any type of prescription or over-the-counter medication, or having any chronic illnesses, which require medical care.
* Inability to complete any of the exercise performance testing on the familiarization day.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-04-15 (Actual)

PRIMARY OUTCOMES:
Symptoms checklist | Change from 0 at 12, 18 and 24 hours
  monitor frequency and severity of subjective symptoms related to a broad spectrum of conditions. The participant is presented with 21 symptoms. The participant is required to rate each symptom (e.g. fatigue, headache, Nausea, numbness/tingling etc. on a scale from 0 (Not Present) to 6 (Severe)
COGcomp (composite measure of cognition) | Change from 0 at 12, 18 and 24 hours
  Throughput (TP) scores from each of seven cognitive assessments administered as part of a battery of tests via Automated Neuropsychological Assessment Metrics (ANAM) computer software. Tests include:
  1. Simple reaction time
  2. Code Substitution
  3. Procedural Reaction Time
  4. Mathematical processing
  5. Matching to sample
  6. Code substitution Delayed
  7. Simple reaction time repeat
Monocyte chemoattractant protein-1 (MCP-1) | Change from 0 at 12, 18 and 24 hours
  Serum concentrations of MCP-1
Macrophage-1-antigen (CD11b) | Change from 0 at 12, 18 and 24 hours
  Surface expression of CD11b on classical monocytes and neutrophils
C-C chemokine receptor 2 (CCR2) | Change from 0 at 12, 18 and 24 hours
  Surface expression of CCR2 on classical monocytes
Interleukin-8 | Change from 0 at 12, 18 and 24 hours
  Serum concentrations of interleukin-8
Lymphocyte function-associated antigen-1 (CD11a) | Change from 0 at 12, 18 and 24 hours
  Surface expression of CD11a on classical monocytes and neutrophils

CONTACTS AND LOCATIONS:
Overall Officials: Adam J Wells, PhD, Principal Investigator — University of Central Florida
Locations (1):
- Kinesiology Research Labs, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No